CLINICAL TRIAL: NCT04146103
Title: Prospective Multicenter Open-label One Arm Trial Investigating a Pumpkin Seed, Isoflavonoid and Cranberry Mix in Lower Urinary Tract Symptoms/Benign Prostatic Hyperplasia
Brief Title: A Pumpkin Seed, Isoflavonoid and Cranberry Mix in LUTS/BPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AJ13
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Novex® made of Pumpkin Seed Extract 550mg, Soy Germ Isoflavonoids 50 mg and Cranberry 50mg. The dose is 2 tablets/day taken orally, for 3 months.
  Interventions: Drug: Novex

INTERVENTIONS:
Drug: Novex — Novex® made of Pumpkin Seed Extract 550mg, Soy Germ Isoflavonoids 50 mg and Cranberry 50mg. The dose is 2 tablets/day taken orally.

SUMMARY:
The aim is to assess the efficacy of a mix of Pumpkin Seed Extract, Soy Germ Isoflavonoids and Cranberry (Novex®) in the management of mild to moderate LUTS in BPH patients. The patients will be evaluated based on the severity of LUTS, urological quality of life, and erectile function.

DETAILED DESCRIPTION:
This is a single-arm prospective open-label trial investigating a combination of pumpkin seed, isoflavonoid and cranberry mix in improving LUTS, urological quality of life, and erectile function in BPH patients. The compound will be administered orally two tablets daily for 3 months. Recruited patients will be seen at 3 visits: initial visit (visit 1), 1-month visit (visit 2) and 3-month visit (visit 3) and their data will be collected in a dedicated case report form.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate LUTS due to BPH for at least 6 months at the initial visit
* no previous therapy or are still symptomatic despite the current use of alpha-blockers

Exclusion Criteria:

* International Prostate Symptom Score (IPSS) > 19
* Prostate cancer
* Urethral stenosis

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
IPSS | At 1 and 3 months visits
  Change in IPSS

SECONDARY OUTCOMES:
IPSS subscores | At 1 and 3 months visits
  Change in IPSS subscores (voiding, filling, nocturia)
uQoL | At 1 and 3 months visits
  Change in uQoL
IIEF-5 | At 1 and 3 months visits
  Change in IIEF-5
Rate of ejaculatory dysfunction and orthostatic hypotension | At 1 and 3 months visits
  Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Elie El Helou, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong WC, Wong EL, Li H, You JH, Ho S, Woo J, Hui E. Isoflavones in treating watchful waiting benign prostate hyperplasia: a double-blinded, randomized controlled trial. J Altern Complement Med. 2012 Jan;18(1):54-60. doi: 10.1089/acm.2010.0077. PMID 22268969
- [Background] Gratzke C, Bachmann A, Descazeaud A, Drake MJ, Madersbacher S, Mamoulakis C, Oelke M, Tikkinen KAO, Gravas S. EAU Guidelines on the Assessment of Non-neurogenic Male Lower Urinary Tract Symptoms including Benign Prostatic Obstruction. Eur Urol. 2015 Jun;67(6):1099-1109. doi: 10.1016/j.eururo.2014.12.038. Epub 2015 Jan 19. PMID 25613154
- [Background] Blanker MH, Bosch JL, Groeneveld FP, Bohnen AM, Prins A, Thomas S, Hop WC. Erectile and ejaculatory dysfunction in a community-based sample of men 50 to 78 years old: prevalence, concern, and relation to sexual activity. Urology. 2001 Apr;57(4):763-8. doi: 10.1016/s0090-4295(00)01091-8. PMID 11306400
- [Background] Kaminetsky J. Comorbid LUTS and erectile dysfunction: optimizing their management. Curr Med Res Opin. 2006 Dec;22(12):2497-506. doi: 10.1185/030079906x154141. PMID 17265598
- [Background] Kaplan SA, DE Rose AF, Kirby RS, O'leary MP, McVary KT. Beneficial effects of extended-release doxazosin and doxazosin standard on sexual health. BJU Int. 2006 Mar;97(3):559-66. doi: 10.1111/j.1464-410X.2005.05959.x. PMID 16469026
- [Background] Damiano R, Cai T, Fornara P, Franzese CA, Leonardi R, Mirone V. The role of Cucurbita pepo in the management of patients affected by lower urinary tract symptoms due to benign prostatic hyperplasia: A narrative review. Arch Ital Urol Androl. 2016 Jul 4;88(2):136-43. doi: 10.4081/aiua.2016.2.136. PMID 27377091
- [Background] Hong H, Kim CS, Maeng S. Effects of pumpkin seed oil and saw palmetto oil in Korean men with symptomatic benign prostatic hyperplasia. Nutr Res Pract. 2009 Winter;3(4):323-7. doi: 10.4162/nrp.2009.3.4.323. Epub 2009 Dec 31. PMID 20098586
- [Background] Vahlensieck W, Theurer C, Pfitzer E, Patz B, Banik N, Engelmann U. Effects of pumpkin seed in men with lower urinary tract symptoms due to benign prostatic hyperplasia in the one-year, randomized, placebo-controlled GRANU study. Urol Int. 2015;94(3):286-95. doi: 10.1159/000362903. Epub 2014 Sep 5. PMID 25196580
- [Background] McMurdo ME, Argo I, Phillips G, Daly F, Davey P. Cranberry or trimethoprim for the prevention of recurrent urinary tract infections? A randomized controlled trial in older women. J Antimicrob Chemother. 2009 Feb;63(2):389-95. doi: 10.1093/jac/dkn489. Epub 2008 Nov 28. PMID 19042940
- [Result] Vidlar A, Student V Jr, Vostalova J, Fromentin E, Roller M, Simanek V, Student V. Cranberry fruit powder (Flowens) improves lower urinary tract symptoms in men: a double-blind, randomized, placebo-controlled study. World J Urol. 2016 Mar;34(3):419-24. doi: 10.1007/s00345-015-1611-7. Epub 2015 Jun 7. PMID 26049866